CLINICAL TRIAL: NCT01607385
Title: A Single Blind, Randomized, Placebo-controlled, Dose Escalating Study to Evaluate the Safety, Tolerability,Pharmacokinetic and Pharmacodynamic Parameters of Repeat Doses of GSK2330672 in Healthy Volunteers, Given Alone and With a Single Day of Dosing With GSK1614235
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetic a Single Day of Dosing With GSK1614235.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116511
Record Dates: First submitted 2012-05-17; First posted 2012-05-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacokinetic; intestinal bile acid transporter inhibitor; GSK2330672; pharmacodynamic; GSK1614235; dose escalation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- GSK2330672 (Active Comparator)
  Interventions: Drug: GSK2330672; Drug: GSK1614235
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: GSK1614235

INTERVENTIONS:
Drug: GSK2330672 — BID, repeat doses
  Arms: GSK2330672
Drug: Placebo — BID, repeat doses
  Arms: Placebo
Drug: GSK1614235 — BID, co-dosed BID with last dosing day of active/placebo repeat doses

SUMMARY:
A single blind, randomized, placebo-controlled, dose escalating study to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic parameters of repeat doses of GSK2330672 in healthy volunteers, given alone and with a single day of dosing with GSK1614235

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Laboratory assessments may be repeated if outside of normal ranges. The Investigator may interpret screening vital sign data based on the subject's age, physical state and level of fitness. Subjects with vital sign readings marginally outside the normal ranges below may be included in the study if in the Investigator's opinion these values are not clinically significant and will not present a safety risk or affect study assessments.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. Subjects must understand the aims, investigational procedures and possible consequences of the study and must be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Male or female between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases, a blood sample with simultaneous follicle stimulating hormone greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 140 pmol/L) is confirmatory in the absence of a clear postmenopausal history; Females on hormone replacement therapy must discontinue hormone replacement therapy to allow confirmation of post-menopausal status prior to study enrollment. For most forms of hormone replacement therapy, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of hormone replacement therapy. Following confirmation of their post-menopausal status, they can resume use of hormone replacement therapy during the study.
* Body mass index within the range 19 - 32kg/m2 (inclusive).

Exclusion Criteria:

* ALT, alkaline phosphatase and bilirubin greater than 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%.
* Current or chronic history of inflammatory bowel disease, chronic diarrhea, Crohn's disease or malabsorption syndromes.
* Current or chronic history of cholelithiasis, inflammatory gall bladder disease, cholestatic liver injury, and cholecystectomy.
* Current or chronic history of liver disease, or known hepatic abnormalities (with the exception of Gilbert's syndrome).
* Fecal occult blood positive test at screening.
* Triglycerides greater than 250mg/dL.
* History of chronic or acute pancreatitis.
* Mean QTc greater than and equal to 450msec on three tracings obtained at least 5 minutes apart.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 14 drinks for males or greater than 7 drinks for females. One drink is equivalent to 12g of alcohol: 12 ounces (360mL) of beer, 5 ounces (150mL) of wine or 1.5 ounces (45mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days or 5 half-lives of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56-day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2012-12-03 (Actual); Study Completion 2012-12-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3 weeks
Clinical laboratory tests for safety. | 7 weeks
  Regular clinical chemistry and hematology panels.
Bristol Stool Form Scale | 2 weeks
  Frequency of bowel movements and quality of stool samples.
Gastrointestinal Symptom Rating Scale | 2 weeks
  Tolerability of possible gastic side effets.

SECONDARY OUTCOMES:
Pharmacokinetic measures of GSK2330672. | Change from baseline at 2 weeks.
  AUC, Cmax, tmax, t1/2
Pharmcokinetic measures of GSK2330672, GSK1614235, GSK2313533, and GSK2313537. | Full profiles on Day 13.
  AUC, Cmax, tmax and t1/2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116511 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116511?search=study&search_terms=116511#rs
- Available data/document: Study Protocol: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116511 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register